CLINICAL TRIAL: NCT03031197
Title: The Supporting Adolescent Adherence in Vietnam (SAAV) Study
Brief Title: Supporting Adolescent Adherence in Vietnam (SAAV)
Acronym: SAAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New England (Other)
Collaborators: Institute of Population, Health and Development, Vietnam (Other); Boston University (Other)
Responsible Party: Principal Investigator, Mary DeSilva, Assistant Research Professor, University of New England
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R21MH109381-01 (NIH)
Record Dates: First submitted 2017-01-21; First posted 2017-01-25 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Adolescents; HIV/AIDS; Patient Adherence
Keywords: adherence; adolescent; HIV/AIDS; Vietnam
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Patient Compliance | interventions — Counseling

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Tailored realtime triggered reminder pkg (Experimental): The core intervention will utilize innovative wireless technology to provide patients with 1) real time, personalized wireless reminder messages when ART doses are not taken on time, and 2) 'feedback' on adherence behavior via monthly interactive counseling sessions informed by summaries of their previous month's behavior. The core intervention will be personalized by each intervention arm patient, who may choose features to suit their preferences.
  Interventions: Combination Product: Tailored realtime triggered reminder pkg
- Control (No Intervention): Comparison subjects will receive usual care and an offer of counseling at monthly clinic visits.

INTERVENTIONS:
Combination Product: Tailored realtime triggered reminder pkg — Core intervention: 1) real time, personalized wireless reminder messages when ART doses are not taken on time, and 2) 'feedback' on adherence behavior via monthly interactive counseling sessions informed by summaries of their previous month's behavior. Personalized features of the intervention will be selected by each patient and may include 1) reminders sent to the WPC (light or chimes) or to patient's or caregiver's cell phone if dose is late; 2) content of text messages from a menu of options; 3) use of "youth-friendly" WPC adherence reports for interactive counseling sessions; 4) additional counseling by clinic staff; 5) a "buddy" system, by choosing someone to review the adherence report with him/her; and 6) a "reward message" after a pre-selected time period of excellent adherence.
  Other Names: wireless monitoring/feedback, counseling, dose histories
  Arms: Tailored realtime triggered reminder pkg

SUMMARY:
The small RCT will assess feasibility, acceptability, and impact of a real-time intervention on ART adherence and clinical outcomes for HIV-positive adolescents. All subjects will use a wireless pill container (WPC) to monitor adherence. Intervention subjects will receive a personalized triggered reminder (cellphone message/call or bottle-based flash/alarm) when they miss a dose, and engage in monthly counseling sessions informed by their adherence data. Comparison subjects will receive usual care and an offer of counseling at monthly clinic visits.

DETAILED DESCRIPTION:
A major priority in HIV care and treatment is identifying effective interventions for adolescent patients, including those that make use of new technologies, to help them achieve and maintain high levels of adherence to antiretroviral treatment (ART), particularly as they take responsibility for their own medication-taking in the transition to adult care. The research planned here will contribute to the scientific evidence base on approaches to support ART adherence effectively among youth by 1) conducting formative research on adherence challenges among adolescents and refining options for a personalized adherence intervention package; and 2) implementing a small randomized controlled trial (RCT) to assess the feasibility, acceptability, and efficacy of a novel real-time feedback intervention that permits adolescent patients to tailor intervention features to suit their individual preferences.

ELIGIBILITY:
Inclusion Criteria:

* currently a patient at the Infectious Disease (ID) clinic at National Hospital for Pediatrics (NHP) in Hanoi, Vietnam
* between 12 and 17 years old of age AND
* expected to remain in care at the NHP for 7 months minimum
* currently on ART
* live in the clinic catchment area
* willing to provide informed assent, caregiver willing to provide consent
* identified ás having adherence challenges (CD4, detectable VL, and/or clinician suggestion)

Exclusion Criteria:

* below the age of 12 years or above the age of 18
* not currently on ART
* live outside the clinic catchment area
* not willing to provide informed assent, caregiver not willing to provide consent

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
Optimal on-time adherence | End of intervention period (month 7)
  Proportion of patients with ≥95% on-time adherence at end of 6-month intervention period in each study arm

SECONDARY OUTCOMES:
CD4 count | Pre-intervention month (month 1) vs. last intervention month (month 7)
  Mean change in CD4 count in each study arm
Viral load | End of intervention period (month 7)
  Percent of patients with undetectable viral load (UDVL) in each study arm

CONTACTS AND LOCATIONS:
Overall Officials: Mary DeSilva, ScD, Principal Investigator — University of New England
Locations (1):
- Institute for Population Health and Development, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided
Undecided.

REFERENCES:
- [Derived] DeSilva M, Vu CN, Bonawitz R, Hai LT, Van Lam N, Yen LT, Gifford AL, Haberer J, Linh DT, Sabin L. The Supporting Adolescent Adherence in Vietnam (SAAV) study: study protocol for a randomized controlled trial assessing an mHealth approach to improving adherence for adolescents living with HIV in Vietnam. Trials. 2019 Feb 28;20(1):150. doi: 10.1186/s13063-019-3239-1. PMID 30819228